CLINICAL TRIAL: NCT05204186
Title: Evaluation of the Impact of COMORBIDities on Morbidity and Mortality After Radical Cystectomy for Cancer Using a Predictive Method With Artificial Intelligence
Brief Title: Impact of COMORBIDities After Radical Cystectomy Using a Predictive Method With Artificial Intelligence
Acronym: COMORBID-AI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0176
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Bladder Cancer; Comorbidity; Deep Learning
Keywords: Bladder Cancer; Comorbidity; Deep learning; PSO-Particle swarm optimization
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patient with (Group A) any Grade 3 (and over) Clavien-Dindo grading complication rate (30dC and 90dC)
- Group B: Patient without (Group B) any Grade 3 (and over) Clavien-Dindo grading complication rate (30dC and 90dC)

SUMMARY:
Clinician and the multidisciplinary team meeting in oncologic urology (MMO) play a key-role in the decision making. An unexplained surgeon attributable variance, probably linked to the subjective "eyeball test" effect, was identified as a strongest factor underlying non-compliance with guide line recommendations in the management of bladder cancer. So high-quality studies that identify barriers and modulators (such as comorbidities) of provider-level adoption of guidelines and how comorbidities are associated in making therapeutic choice and their impact in bladder cancer specific survival and overall survival, are crucial. To identify patients at high risk of early death, and to improve specific guideline for treatment might be decisive.

In order to assess survival, where mortality events compete, it will be more appropriate to compute a Cumulative Incidence Function (namely CIF). The investigators will compare outcomes across patient populations to obtain information to improve clinical decision-making. Such learning will be done through the use of neural networks or by applying population-based approaches, such as Genetic Algorithms (GA), Ant Colony Systems (ACS) and Particle Swarm Optimization (PSO), using as a four-stage based approach.

First, the investigators propose a "pretopology space" in order to study a dynamic phenomenon. Second, the investigators recall that the K-means approach remains one of the most used approaches for classifying a set of elements (patients / persons / others) into K (disjunctive) clusters. Third, the investigators propose a learning pretopology space for enhancing the clustering. Such an approach can be assimilated in spirit to one applied with high success on deep learning. Fourth and last, the investigators propose a reactive method that is able to include some new elements or remove some contained elements

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patient treated by radical cystectomy for bladder cancer

Exclusion Criteria:

* Computed tomography/magnetic resonance evidence of distant metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective analysis of data from patients treated by radical cystectomy in our institution from 01 January 2006 to 01 January 2021. Qualitative and quantitative standard tumour data elements will be retrieved from medical files and certified General Cancer Registry. Data collection will be conducted from 9/2021 to 9/2022. Data management and analysis will be conducted from 1/2023 to 12/2024.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
bladder cancer therapeutic choice as determined with this Artificial Intelligence predictive method | 90 days
  After retrieving associated comorbidities, any Grade 3, and over, Clavien-Dindo grading system complication rate (30dC and 90dC), information on primary treatment for bladder cancer (urothelial type and pT1 to pT4), outcome, time and cause of death, by our technician (from medical files of specific support centers), the primary objectives will be to model incorporation of comorbidities in making therapeutic choice, to improve care for patients with bladder cancer and specific guideline for treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No